CLINICAL TRIAL: NCT01793753
Title: Effect of Propofol on Internal Anal Sphincter Pressure During ARM
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jaime Belkind-Gerson, MD, Medical Director, Neurogastroenterology, Massachusetts General Hospital
Other Study IDs: 2012P000231
Record Dates: First submitted 2013-02-05; First posted 2013-02-18 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Propofol: Chronically constipated children ages 2-6 years who will receive anesthesia for anorectal manometry including propofol per standard of care
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol

SUMMARY:
Background and Aim: An anorectal manometry (ARM) is a common test in the evaluation of outlet obstruction in constipation. In children under 6 yo, anesthesia is often used for patient comfort and compliance. The choice of anesthesia for ARM varies from center to center and includes the use of ketamine, inhalation agents, and propofol. With the increased use of propofol, our aim is to determine the effects of propofol on resting anal sphincter pressure while performing an ARM under general anesthesia.

Hypothesis: Propofol administration leads to a decrease in internal anal sphincter pressure.

Methods: This is a prospective, single center, observational study of the effect of propofol on the internal anal sphincter pressure. Pediatric patients between the ages of 2-6 years who require an anorectal manometry for chronic constipation will be offered enrollment. Anesthesia was required for patient compliance and comfort and conducted by an anesthesiologist. Sevoflurane was the inhalational agent used for induction. At Massachusetts General Hospital (MGH), 1 mg/kg of propofol bolus is routinely given at completion of the ARM test to reduce emergence delirium. The manometric probe was kept in place with continuous measurement of baseline internal anal sphincter pressure while propofol was administered. We measured changes to internal anal sphincter pressure and time to return to baseline.

Results: The primary outcomes will be change of internal anal sphincter pressure from baseline and time to return to baseline.

Discussion: The proposed investigation may demonstrate that propofol has an effect on the internal anal sphincter pressure which may affect its utility as an anesthetic for anorectal manometry.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 - 6 years
* Chronic constipation
* Requires anorectal manometry

Exclusion Criteria:

* Ages 0-2 or > 6 years
* Abnormal anorectal anatomy
* Known history of Hirschsprung's Disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Chronically constipated children ages 2-6 years who will receive anesthesia for anorectal manometry including propofol per standard of care
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in internal anal sphincter pressure from baseline | Patients will be followed for the duration of outpatient anal rectal manometry procedure, an average of 10 minutes
  Baseline internal anal sphincter pressures will be measured at start of anorectal manometry. Patients will be followed for the duration of the procedure (~10 minutes). After propofol is given at end of procedure, changes to baseline internal anal sphincter pressure will be measured until return to baseline (up to 5 minutes)
Time for internal anal sphincter pressure to return to baseline | Patients will be followed for the duration of outpatient anal rectal manometry procedure, an average of 10 minutes
  Patients will be followed for the duration of the procedure (~10 minutes). After propofol is given at end of procedure, changes to baseline internal anal sphincter pressure will be measured until return to baseline (up to 5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Belkind-Gerson, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tran K, Kuo B, Zibaitis A, Bhattacharya S, Cote C, Belkind-Gerson J. Effect of propofol on anal sphincter pressure during anorectal manometry. J Pediatr Gastroenterol Nutr. 2014 Apr;58(4):495-7. doi: 10.1097/MPG.0000000000000190. PMID 24121151